CLINICAL TRIAL: NCT03274544
Title: The Effectiveness of an Empirical Chinese Medicine Formulation for Idiopathic Pulmonary Fibrosis: an Open Label Clinical Trial
Brief Title: Clinical Trial of Chinese Herbal Medicine for Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting eligible patients
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, Associate Director (Clinical Affairs), The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 17-283
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Chinese Medicine; Herbal Medicine
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROLUNG (Experimental): Herbal formula treatment PROLUNG in additional to current therapy
  Interventions: Other: PROLUNG

INTERVENTIONS:
Other: PROLUNG — Chinese herbal medicine formula PROLUNG with individual herbs of the formula are listed as follows (weight in granule preparation):
  * Huang Qi (Radix Astragali Membranaceus): 2 g
  * Dan Shen (Radix Salviae Miltiorrhizae): 1 g
  * Jiang Huang (Rhizoma Curcumae Longae): 1 g
  * Yin Xing (Semen Gingko Bilobae): 1 g
  * Mai Men Dong (Tuber Ophiopogonis Japonoci): 1 g
  * Bai He (Bulbus Lilii): 1g
  * Jin Yin Hua (Flos Lonicerae Japonicae): 1 g
  * Zi Su Ye (Folium Perillae Frutescentis): 1 g
  * Yin Yang Huo (Herba Epimedii): 1g

SUMMARY:
This open label clinical study will be conducted in School of Chinese Medicine Clinics at The University of Hong Kong (HKU) to preliminarily determine whether treatment with the herbal formula PROLUNG could improve Idiopathic Pulmonary Fibrosis (IPF) symptoms, respiratory function and the quality of life of patients with IPF compared with pretreatment baseline. We propose to recruit 30 participants. The diagnosis and screening will be conducted by respiratory physicians. Those who meet the inclusion criteria will be referred by the expert to the PI. The PI will prescribe the formula in granule form to the participants in Traditional Chinese medicine (TCM) Clinics as usual. Patients will receive 6 months of the herbal treatment and 7 visits.

Annual rate of change in forced expiratory vital capacity (FVC) will serve the primary outcome. The St. George's Respiratory Questionnaire (SGRQ) will be used to additionally assess respiratory functions. A standard questionnaire will be administered to obtain information on age, sex, marital status, education, social class, smoking behaviour and respiratory diseases. Other outcome measures include the 36-Item Short Form Survey (SF-36) and the World Health Organization Quality of Life assessment instrument (WHOQOLBREF) by each participant after enrollment.

DETAILED DESCRIPTION:
Background Idiopathic pulmonary fibrosis (IPF) is a dreadful disease characterized by progressive impairment in quality of life, increasingly limited physical function, and an early death from respiratory failure. IPF is the most common and predominantly lethal form of the idiopathic interstitial pneumonias, with an associated median survival of only 2 to 3 years. The etiology of this chronic and progressive fibrotic lung disease is unknown, although potential risk factors such as cigarette smoking and other environmental exposures have been described. In a study published in 2006 based on a United States healthcare claims database, the prevalence of IPF was between 14-42.7 per 100,000, depending on whether narrow or broad case-finding criteria was used. IPF is more commonly seen in patients between 40 to 70 years of age. The risk of death as a result of IPF also increases with age, with a hazard ratio of 0.25 for patients younger than 50 years and a longer median survival amongst those younger than 50 (116.4 months compared to 62.8 months). IPF occurs more commonly in men than in women and also progress faster and result in worse survival in men. The IPF mortality rate in the United States was found to be 61.2 deaths per 1,000,000 in men and 54.5 per 1,000,000 in women, nevertheless, the death rate in women is increasing at a faster rate than in men. Age-adjusted mortality has been found to be greater among whites than blacks and is increasing at a higher rate among whites when compared to other racial and ethnic groups. There is no effective treatment for IPF, although pirfenidone and nintedanib have been approved for treatment of IPF, with benefit in slowing down lung function decline. At present, the only intervention that improves survival in select patients with IPF is lung transplantation. With this to look forward to, it is no surprise that patients and their physicians are desperate for treatment options that might change the outcome. Traditional Chinese herbal medicine has been an important source to treat this ailment.

Traditional Chinese medicine (TCM) has dealt with IPF for long time. A condition similar to pulmonary fibrosis can be found in Chinese literature thousands years ago. A disease termed "Fei Wei" was described and is similar to IPF in definition, pathophysiology, and treatment. It was reported that the disease was extremely difficult to treat. Other TCM terms of respiratory disease similar to IPF were "short breath", "cough", "lung inflation", and "Fei Bi".

In recent years, TCM has renewed its focus on pulmonary fibrosis and other respiratory illnesses because of SARS (Severe Acute Respiratory Syndrome), a viral infection which spread in China in late 2002 and 2003. SARS infection resulted in pulmonary fibrosis in a number of individuals who contracted SARS, although the pathophysiology of pulmonary fibrosis resulting from SARS may differ from that of IPF, the fibrosis can be reversible. In TCM, the pathophysiology for IPF is a complex of group of terms: Feng (Wind-external factor), Re (Heat-inflammation), Tan (Phlegm), Yu (Congestion). Treatment may vary according to the phases of the disease, symptoms, and individuals.

IPF causes pulmonary interstitial chronic inflammation, immune complex deposition in the lung interstitium into fibroblasts and collagen eventually leads to the destruction of lung tissue. In TCM terms, this represents Blockage of Heat in the lung. With Heat in the pulmonary mass, the Lung loses the function of controlling Qi, hence the patients suffers difficulty in breathing, has no air suction, has shortness of breath, dry cough, wheezing, and other symptoms.

In China, herbal medicine is the main treatment for IPF. Research has shown the effectiveness of traditional Chinese herbs formulations developed to treat IPF. The Individual herbs of the formula have been widely used to improve pulmonary function.

Current evidence Chinese herbal medicine formula used in the proposed study

Our empirical evidence suggests that one Chinese herbal medicine formula PROLUNG has considerable benefit in the treatment of IPF. Individual herbs of the formula are listed as follows (weight in granule preparation):

Huang Qi (Radix Astragali Membranaceus): 2 g Dan Shen (Radix Salviae Miltiorrhizae): 1 g Jiang Huang (Rhizoma Curcumae Longae): 1 g Yin Xing (Semen Gingko Bilobae): 1 g Mai Men Dong (Tuber Ophiopogonis Japonoci): 1 g Bai He (Bulbus Lilii): 1g Jin Yin Hua (Flos Lonicerae Japonicae): 1 g Zi Su Ye (Folium Perillae Frutescentis): 1 g Yin Yang Huo (Herba Epimedii): 1g

The therapeutic effects in treating IPF: One study in animal model of IPF has shown that treatment with an herbal formula including Ginseng, Mai Men Dong, Tao Ren, Chi Shao, Neu Xi, Jie Geng, Dang Gui, Di Hung, Ban Xia, Gan Cao, Zhi Ke, and Hong Hua inhibited B cell hyperactivity, which may be related to fibrosis. IPF patients treated with a combination of traditional Chinese herbs and drugs improve faster and remain free of IPF longer than patients treated with drugs alone. One 2-month study was performed in 12 patients with IPF to find out the effect of a combination of Dang Shen, Huang Qi, Sha Shen, Mai Men Dong, Dang Gui, Dan Shen, Chuan Xiong, Sang Bei Pi, Xing Ren, Bai Guo, Huang Qin, Ban Xia, Ma Huang, and Gan Cao. The patients were exclusively provided with the Chinese herb formulation except when the illness worsened. The results have shown an improvement in dyspnea and cyanosis and an increase in PO2 (partial pressure of oxygen) in 5 of the 12 patients.

Dan Shen (Radix Salviae Miltiorrhizae): Dan Shen and its purified active component IH764-3, have been shown to prevent pulmonary fibrosis induced with bleomycin. The Chinese herb formulation blocks the expression of TGF-alpha1 and inhibits the activity of fibroblast growth factor when administered 24 hours after bleomycin-induction. Dan Shen has also been used successfully in the treatment of allergic rhinitis by bilateral injection into the inferior nasal choncha.

Huang Qi (Radix Astragali Membranaceus): Astragaloside is the main ingredient in Huang Qi, and is known to have antiinflammatory, anti-fibrotic, and immunoregulatory properties. It was reported to improve lung functions in mice experimentally induced chronic asthma by reducing the amount of hydroxyproline, an indicator of pulmonary fibrotic activity. The administration of Huang Qi in a population with history of bronchial asthma, allergic rhinitis, and chronic bronchitis, Huang Qi prevents against pulmonary tract infections. Among 30 patients with IPF treated with Huang Qi in combination with other Chinese herb formulations, 3.87% showed larger increase in diffusing capacity of the lung for carbon monoxide (DLCO) as compared with patients treated with prednisone in a clinical study. A combination of Huang Qi, Dan Shen and prednisone was given to 19 patients who had a 3.75% greater improvement in total lung capacity, a 4.01% greater improvement in vital capacity, and a 3.78% greater increase in DLCO than 19 other patients who exclusively received prednisone. Dan Shen and Huang Qi were components in an herbal combination that resulted in 3- and 5- year survival rates in subjects with IPF.

Jiang Huang (Rhizoma Curcumae Longae): Jiang Huang's anti-inflammatory properties have been established in rats. Curcumin, which is derived from Jiang Huang, also has anti-carcinogenic and antioxidant characteristics. Curcumin can limit the expression of tumor growth factor- β (TGF-β). It can also reduce TGF-β signaling in renal fibroblasts in vitro. It has been shown to limit hydroxyproline levels in the lungs of mice exposed to bleomycin and to prevent alveolitis in mice with bleomycin-induced IPF.

Yin Xing (Semen Gingko Bilobae): Yin Xing is recommended to treat chronic cough, asthma, chronic wheezing, phlegm, and chronic voice loss. The bronchodilation and expectorant properties of Yin Xing have been established.

Mai Men Dong (Tuber Ophiopogonis Japonoci): For chronic dry cough and sore throat, Mai Men Dong is a recommended treatment. Mai Men Dong in combination with other traditional Chinese herbs was shown to be effective in the treatment of allergic asthma in children.

Bai He (Bulbus Lilii): Bai He is recommended to be used in combination with other herbs, in the treatment of dry cough, bronchiectasis, and hemoptysis and alone in the treatment of lung abcesses.

Jin Yin Hua (Flos Lonicerae Japonicae): Jin Yin Hua is recommended to treat pneumonia, bronchitis, and upper respiratory tract infections in general in combination with other herbs.

Zi Su Ye (Folium Perillae Frutescentis): Zi Su Ye improves bronchodilation, decreases bronchioli excretions and relieves bronchiospasms.

Yin Yang Huo (Herba Epimedii): Yin Yang Huo has expectorant, antiasthmatic, and antitussive actions. Yin Yang Huo has shown effectiveness to treat chronic bronchitis.

Toxic profiles and herb interactions: Individual herbs used in the formula are in general safe and well tolerated within therapeutic doses. Dan Shen increased the effect of warfarin when the two medications are taken together. Dan Shen also increased the activity of liver enzymes involved in drug metabolism, thereby increasing drug metabolism rates. Jiang Huang may also exacerbate the effects of warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Either gender aged 40-75;
* Has a diagnosis of IPF, made by a respiratory expert based on International Classification of Diseases (ICD-10);
* No participation in another clinical study within 4 weeks of study start.
* Participation in this study must be voluntary and not coerced.

Exclusion Criteria:

* Have received lung transplantation.
* Any condition that may compromise patient safety.
* Pregnant women or women trying to become pregnant will be excluded from the study.
* History of drug or alcohol abuse within 6 months of study start.
* History of immunocompromise, including a positive HIV test result.
* Impaired liver and renal functions.
* Known allergies to any Chinese herbs and participants with numerous or severe allergies to any allergen.
* Pre-existing conditions including renal failure, chronic renal problems, chronic hepatitis, other pulmonary problems, diabetes, and heart problems will be excluded from the study.
* Either mentally incompetent or are unable to give informed consent because of the language barrier.
* Taking the following drugs, even as part of their current treatment regimen for IPF: pirfenidone, nintedanib, antiplatelet drugs (including aspirin, clopidogrel (Plavix), and dipyridamole (Persantine), anticoagulant drugs (including warfarin (Coumadin), enoxparin (Lovenox), and heparin), cardiac glycosides (e.g. digoxin), sedatives and sedative-containing drugs (including barbiturates, narcotic analgesics, benzodiazepines, and antihistamines), and traditional Chinese herbal medicines or granules, or other herbal medicines or supplements.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Annual rate of change in forced expiratory vital capacity (FVC) | Baseline, 6 month
  Annual rate of change in forced expiratory vital capacity (FVC) will serve the primary outcome.

SECONDARY OUTCOMES:
Changes in SGRQ score | Baseline, 1 month, 2 month, 3 month, 4 month, 5 month, 6 month
  The St. George's Respiratory Questionnaire (SGRQ) will be used to additionally assess respiratory functions.
Changes in SF-36 score | Baseline, 1 month, 2 month, 3 month, 4 month, 5 month, 6 month
  The 36-Item Short Form Survey (SF-36) is a 36-question questionnaire to assess the quality of life of a participant in terms of physical and mental health.
Changes in WHOQOL-BREF score | Baseline, 1 month, 2 month, 3 month, 4 month, 5 month, 6 month
  The WHOQOL-BREF measures the physical and psychological health, the social relationships, and the environment of an individual.
Changes in adverse events | Baseline, 1 month, 2 month, 3 month, 4 month, 5 month, 6 month
  All patients will be monitored for adverse reactions of any kind including but not limited to idiosyncratic allergic reactions to some components of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin ZHANG, MMed, PhD, Principal Investigator — zhangzj@hku.hk
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Raghu G, Weycker D, Edelsberg J, Bradford WZ, Oster G. Incidence and prevalence of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2006 Oct 1;174(7):810-6. doi: 10.1164/rccm.200602-163OC. Epub 2006 Jun 29. PMID 16809633
- [Background] Navaratnam V, Fleming KM, West J, Smith CJ, Jenkins RG, Fogarty A, Hubbard RB. The rising incidence of idiopathic pulmonary fibrosis in the U.K. Thorax. 2011 Jun;66(6):462-7. doi: 10.1136/thx.2010.148031. Epub 2011 Apr 27. PMID 21525528
- [Background] Erbes R, Schaberg T, Loddenkemper R. Lung function tests in patients with idiopathic pulmonary fibrosis. Are they helpful for predicting outcome? Chest. 1997 Jan;111(1):51-7. doi: 10.1378/chest.111.1.51. PMID 8995992
- [Background] King TE Jr, Tooze JA, Schwarz MI, Brown KR, Cherniack RM. Predicting survival in idiopathic pulmonary fibrosis: scoring system and survival model. Am J Respir Crit Care Med. 2001 Oct 1;164(7):1171-81. doi: 10.1164/ajrccm.164.7.2003140. PMID 11673205
- [Background] Han MK, Murray S, Fell CD, Flaherty KR, Toews GB, Myers J, Colby TV, Travis WD, Kazerooni EA, Gross BH, Martinez FJ. Sex differences in physiological progression of idiopathic pulmonary fibrosis. Eur Respir J. 2008 Jun;31(6):1183-8. doi: 10.1183/09031936.00165207. Epub 2008 Mar 5. PMID 18321929
- [Background] Gribbin J, Hubbard RB, Le Jeune I, Smith CJ, West J, Tata LJ. Incidence and mortality of idiopathic pulmonary fibrosis and sarcoidosis in the UK. Thorax. 2006 Nov;61(11):980-5. doi: 10.1136/thx.2006.062836. Epub 2006 Jul 14. PMID 16844727
- [Background] Olson AL, Swigris JJ, Lezotte DC, Norris JM, Wilson CG, Brown KK. Mortality from pulmonary fibrosis increased in the United States from 1992 to 2003. Am J Respir Crit Care Med. 2007 Aug 1;176(3):277-84. doi: 10.1164/rccm.200701-044OC. Epub 2007 May 3. PMID 17478620
- [Background] Rafii R, Juarez MM, Albertson TE, Chan AL. A review of current and novel therapies for idiopathic pulmonary fibrosis. J Thorac Dis. 2013 Feb;5(1):48-73. doi: 10.3978/j.issn.2072-1439.2012.12.07. PMID 23372951
- [Background] Antonio GE, Wong KT, Hui DS, Wu A, Lee N, Yuen EH, Leung CB, Rainer TH, Cameron P, Chung SS, Sung JJ, Ahuja AT. Thin-section CT in patients with severe acute respiratory syndrome following hospital discharge: preliminary experience. Radiology. 2003 Sep;228(3):810-5. doi: 10.1148/radiol.2283030726. Epub 2003 Jun 12. PMID 12805557
- [Background] Chan KS, Zheng JP, Mok YW, Li YM, Liu YN, Chu CM, Ip MS. SARS: prognosis, outcome and sequelae. Respirology. 2003 Nov;8 Suppl(Suppl 1):S36-40. doi: 10.1046/j.1440-1843.2003.00522.x. PMID 15018132
- [Background] Xie L, Liu Y, Fan B, Xiao Y, Tian Q, Chen L, Zhao H, Chen W. Dynamic changes of serum SARS-coronavirus IgG, pulmonary function and radiography in patients recovering from SARS after hospital discharge. Respir Res. 2005 Jan 8;6(1):5. doi: 10.1186/1465-9921-6-5. PMID 15638943
- [Background] Yang J, Cui Y, Kolb M. How useful is traditional herbal medicine for pulmonary fibrosis? Respirology. 2009 Nov;14(8):1082-91. doi: 10.1111/j.1440-1843.2009.01644.x. PMID 19909458
- [Background] Hsu CH, Lu CM, Chang TT. Efficacy and safety of modified Mai-Men-Dong-Tang for treatment of allergic asthma. Pediatr Allergy Immunol. 2005 Feb;16(1):76-81. doi: 10.1111/j.1399-3038.2005.00230.x. PMID 15693916
- [Background] Zhou L, Zuo Z, Chow MS. Danshen: an overview of its chemistry, pharmacology, pharmacokinetics, and clinical use. J Clin Pharmacol. 2005 Dec;45(12):1345-59. doi: 10.1177/0091270005282630. PMID 16291709
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Background] Kalantar-Zadeh K, Kopple JD, Block G, Humphreys MH. Association among SF36 quality of life measures and nutrition, hospitalization, and mortality in hemodialysis. J Am Soc Nephrol. 2001 Dec;12(12):2797-2806. doi: 10.1681/ASN.V12122797. PMID 11729250
- [Background] Yao CF, Jiang SL. [Prevention and treatment of pulmonary-fibrosis by traditional Chinese medicine]. Zhong Xi Yi Jie He Xue Bao. 2003 Sep;1(3):234-8. doi: 10.3736/jcim20030327. Chinese. PMID 15339572
- [Background] Costabel U, King TE. International consensus statement on idiopathic pulmonary fibrosis. Eur Respir J. 2001 Feb;17(2):163-7. doi: 10.1183/09031936.01.17201630. No abstract available. PMID 11334114
- [Background] Mannino DM, Etzel RA, Parrish RG. Pulmonary fibrosis deaths in the United States, 1979-1991. An analysis of multiple-cause mortality data. Am J Respir Crit Care Med. 1996 May;153(5):1548-52. doi: 10.1164/ajrccm.153.5.8630600.
- [Background] Jin Gui Yao Lue (Essentials from the Golden Cabinet), written by Zhang Zhong-jing (about 150-219) in Later Han Dynasty.
- [Background] Huangdi Neijing (The Book of Yellow Emperor's: a classic of internal medicine) written during the period 475-225 b.C. as a dialogue between the mythical Emperor Huangdi and his physician Qibo.
- [Background] Tang ling Hua, Li Chun sheng. special onset of diffuse interstitial pulmonary fibrosis treated 13 cases reported. Traditional Chinese Medicine, 1997, 38 (1): 34 ~ 36.
- [Background] Zhang. L. 1999. A Case Report on Chronic Lymphocytic Leukemia. Journal of Traditional Chinese Medicine Alumni 1: 15.
- [Background] Chen, J.K., Chen, T.T. 2004. Chinese Medical Herbology and Pharmacology. City of Industry, CA: Art of Medicine Press, Inc. 1267pp.
- [Background] Fruehauf, H. 1997. The Gingko. Cultural Background and Medicinal Usage in China. Journal of Chinese Medicine 55: 13-16.
- [Background] Bensky, D., Clavey, S., Stöger, E. 2004. Chinese Herbal Medicine Materia Medica, 3rd Edition. Seattle: Eastland Press, Inc. 1311pp.
- [Background] World Health Organization 1993. WHOQoL Study Protocol. WHO (MNH7PSF/93.9).
- [Background] World Health Organization. 2004. WHO Quality of Life-BREF (WHOQOL-BREF). http://www.who.int/substance_abuse/research_tools/whoqolbref/en/, http://www.who.int/substance_abuse/research_tools/en/english_whoqol.pdf Accessed 09 April 2011.
- [Background] Murphy, B., Herrman, H., Hawthorne, G., Pinzone, T., Evert, H. 2000. Australian WHOQoL instruments: User's manual and interpretation guide. Australian WHOQoL Field Study Centre, Melbourne, Australia.